CLINICAL TRIAL: NCT02632981
Title: IL-32 Levels in Gingival Crevicular Fluid and Saliva of Patients With Chronic Periodontitis After Periodontal Treatment.
Brief Title: IL-32 Levels in Patients With Chronic Periodontitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Figen ÖNGÖZ DEDE, Bülent Ecevit University Faculty of Dentistry, Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 2014-10-14-01
Record Dates: First submitted 2015-12-10; First posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Periodontitis
Keywords: Interleukin-32; periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- chronic periodontitis patients (Active Comparator): gingival crevicular fluid and saliva collecion were taken before and after nonsurgical periodontal treatment
  Interventions: Other: nonsurgical periodontal treatment
- periodontally healthy controls (Placebo Comparator): gingival crevicular fluid and saliva collection were taken at baseline after oral hygiene instructions
  Interventions: Other: Gingival crevicular fluid and saliva collection

INTERVENTIONS:
Other: nonsurgical periodontal treatment — Scaling and root planning under local anaesthesia, in a total of four clinical visits Oral hygiene instructions including the modified Bass technique, regular toothpaste, and an appropriate interdental cleaning device with dental floss and interdental brush.
  Other Names: chronic periodontitis patients
  Arms: chronic periodontitis patients
Other: Gingival crevicular fluid and saliva collection — GCF collection with filter paper (Periopaper) using the intracrevicular method. Patients' mouths were rinsed with distilled water, and unstimulated salivary samples were collected by patients expectorating into disposable tubes.
  Other Names: periodontally healthy controls; chronic periodontitis patients
  Arms: periodontally healthy controls

SUMMARY:
Interleukin-32 (IL-32) is a recently described cytokine that is a strong inducer of pro-inflammatory cytokines such as tumor necrosis factor (TNF)-α. A previous report have reported that Porphyromonas gingivalis-derived LPS significantly up-regulated IL-32 expression compared with the unstimulated cells in monocytes (THP-1 cells). They suggested that IL-32 may contribute to the pathogenesis of periodontal disease. In the present study the investigators hypothesized that IL-32 levels may increase in the gingival crevicular fluid (GCF) and saliva of patients with chronic periodontitis compared with healthy controls and these levels may decrease together with treatment.

DETAILED DESCRIPTION:
The purpose of this study was to investigate IL-32 levels in the GCF and saliva of patients with chronic periodontitis and to evaluate changes after nonsurgical periodontal therapy.

Twenty-seven CP and 27 periodontally healthy controls were enrolled in this study. Periodontitis patients received nonsurgical periodontal treatment. GCF and saliva sampling and clinical periodontal parameters were assessed before and a month after treatment. IL-32, IL-10 and TNF-α levels in GCF and saliva were measured by enzyme-linked immunosorbent assay.

Unstimulated salivary samples were collected using standard techniques. About 2 mL whole saliva was collected in disposable tubes and centrifuged immediately to remove cell debris (10,000 g x 10 minutes). The supernatants (50µL each) were stored at -40C until analyzed. GCF samples were collected from a mesio-buccal and disto-palatal site on each tooth. In the CP group, the samples were obtained from patients at areas with ≥5 mm CAL, ≥6 mm PD and ≥30% bone loss. In the healthy group, GCF samples were collected from teeth exhibiting PD<3 mm without CAL and BOP. The area was isolated with cotton rolls, saliva contamination elimination was ensured, and it was slightly air dried. GCF was sampled with paper strips. Paper strips were placed into the crevice until mild resistance was felt (intracrevicular method) and left in the position for 30 seconds. Strips contaminated with blood or saliva were discarded. Each sampled strip was placed into a 400µl eppendorf centrifuge tube and stored at -40C until analyzed.

ELIGIBILITY:
Inclusion Criteria:

* all subjects in the study were possess of at least 20 teeth excluding third molars.

Exclusion Criteria:

* agressive periodontitis,
* periapical pathologies,
* excessive forces including mechanical forces caused by orthodontic forces and occlusal forces;
* presence of systemic diseases;
* administration of non-steroidal and anti-inflammatory drugs or antibiotic therapies within the previous 6 months;
* need for antibiotic prophylaxis for dental treatment and having received non-surgical periodontal treatment within the past 6 months or surgical periodontal treatment within the past 12 months;
* allergy or sensitivity to any drug,
* pregnancy,
* lactation, and
* current and former use of tobacco.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Biochemical parameters (IL-32, IL-10 and THF-alpha) | Baseline and 1 month after treatment
  The changes in levels of IL-32 after periodontal treatment determined by ELISA. The changes in levels of IL-32 were analyzed to determine diagnostic and prognostic potential as a biomarker of periodontitis.

SECONDARY OUTCOMES:
Probing pocket depth | Baseline and 1 month after treatment
  The changes in probing pocket depth after periodontal treatment.Probing pocket depth was measured for determining severity of disease and clinic outcome.
Probing pocket depth and clinical attachment level | Baseline and 1 month after treatment
  The changes in clinical attachment level after periodontal treatment. The probing depth and the distance from the gingival margin to the cemento-enamel junction are used to measurement of clinical attachment level. Clinical attachment level was measured for determining severity of disease and clinic outcome.
Gingival index | Baseline and 1 month after treatment
  The changes in gingival index after periodontal treatment. Gingival index was recorded for classifying and evaluating (coronally) gingival inflammation.
Plaque index | Baseline and 1 month after treatment
  The changes in plaque index after periodontal treatment. Plaque index was recorded for determining and classifying oral hygiene status.
Bleeding on probing | Baseline and 1 month after treatment
  The changes in bleeding on probing after periodontal treatment. Bleeding on probing was recorded for classifying and evaluating (apically) gingival inflammation.